CLINICAL TRIAL: NCT06581029
Title: Evaluating Mental Health Challenges in Juvenile Lupus Erythematosus and Their Caregivers
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sahar Samir Farghly Badran, pediatric resident, Assiut University
Other Study IDs: J.SLE and psychiatry
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-08

CONDITIONS: SLE

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control healthy group: is 1) no history of psychiatric and medical disease 2) Intelligence quotation more than 70.
- SLE group: I. Age from 11 to 18 years II. Both sex III. diagnosed with SLE for at least 6 months to allow for an adjustment period following diagnosis.
  use of The multidimensional peer victimization scale (PVS), a self-report scale for children and adolescents, was used to assess the victimization
  Interventions: Other: The multidimensional peer victimization scale (PVS)

INTERVENTIONS:
Other: The multidimensional peer victimization scale (PVS) — The multidimensional peer victimization scale (PVS), a self-report scale for children and adolescents, was used to assess the victimization
  Groups: SLE group

SUMMARY:
assessment of psychiatric problems in pediatric SLE and their caregivers. evaluate the possible risk factors of psychiatric problems such as peer victimization, academic performance, fatigue, self-esteem and quality of life.

DETAILED DESCRIPTION:
Juvenile-onset systemic lupus erythematosus (jSLE) is a rare but severe multisystem autoimmune disease which may cause significant damage, disability, and death . Juvenile SLE patients constitute 15-20% of all SLE cases . Compared to the adult SLE, jSLE patients have higher morbidity and mortality rates. Renal, cardiovascular, and neuropsychiatric (NP) involvements are the most important reasons for morbidity and mortality .

Therefore, knowledge of common mental illnesses such as major depressive disorder (MDD) and anxiety disorders in cSLE may be limited. Establishing the prevalence of MDD and anxiety in cSLE is important , as comorbidity rates of these disorders may be increased in cSLE for several reasons. First, the diagnosis of a serious physical health condition confers psychological vulnerability to feelings of sadness, helplessness, stress, and worry about the future.9 For some individuals, such symptoms warrant further evaluation and may persist beyond the initial adjustment period and reach clinical significance, requiring therapeutic intervention. SLE carries a patient-treatment burden similar to other chronic diseases. Such treatment burden places susceptible individuals at risk of psychiatric disorder. Second, although depressed mood may present in the absence of active CNS disease, it may also occur as a symptom of neuropsychiatric c SLE (NPSLE), yielding clinically significant treatment implications. Third, treatment of SLE with known depressogenic medications like steroid may lead to depressive symptom elevation or exacerbate a co-morbid primary MDD. Moreover, among patients with depressed mood as a manifestation of NPSLE, the initiation of steroid treatment may worsen depressive symptoms. It is unclear whether such risks are observed in the cSLE population.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 11 to 18 years
2. Both sex
3. diagnosed with SLE for at least 6 months to allow for an adjustment period following diagnosis.
4. Met the New ACR and EULAR criteria for classification of SLE .

Inclusion criteria of the control healthy group : 1- no history of psychiatric and medical disease 2-Intelligence quotation more than 70.

Exclusion Criteria:

1. No history of psychiatric illness prior to the diagnosis of lupus.
2. Intelligence quotation more than 70.

Ages: 11 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: : this study will include patients who already diagnosed with SLE and following in allergy&immunology and rheumatology unit assiut university children hospital
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluating mental health challenges in juvenile SLE and their caregivers | baseline
  The aim of the present study is to evaluate and assess psychiatric problems in juvenile systemic lupus erythematosus patients and their caregivers. Also, to evaluate the possible risk factors of psychiatric problems such as peer victimization, academic performance, fatigue, self-esteem and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Ali, Professor of pediatric, Study Director — Assiut University; Gellan Karamallah Ramadan Ahmed, lecturer of psychiatry, Study Director — Assiut University; Naglaa Samy, Associate proff, Study Director — Assiut University

REFERENCES:
- [Background] Sarwar S, Mohamed AS, Rogers S, Sarmast ST, Kataria S, Mohamed KH, Khalid MZ, Saeeduddin MO, Shiza ST, Ahmad S, Awais A, Singh R. Neuropsychiatric Systemic Lupus Erythematosus: A 2021 Update on Diagnosis, Management, and Current Challenges. Cureus. 2021 Sep 14;13(9):e17969. doi: 10.7759/cureus.17969. eCollection 2021 Sep. PMID 34667659
- [Background] The American College of Rheumatology nomenclature and case definitions for neuropsychiatric lupus syndromes. Arthritis Rheum. 1999 Apr;42(4):599-608. doi: 10.1002/1529-0131(199904)42:43.0.CO;2-F. PMID 10211873
- [Background] Ho RC, Mak A. The interface between medicine and psychiatry: neuropsychiatric aspects of systemic lupus erythematosus (SLE). Ann Acad Med Singap. 2014 Aug;43(8):388-90. No abstract available. PMID 25244986